CLINICAL TRIAL: NCT00933218
Title: Effects of Polyphenols on Changes of Inflammatory and Cardiovascular Status After a Marathon Run
Brief Title: Beer, Marathon, Genetics, Inflammation and the Cardiovascular System: Be-MaGIC-Trial
Acronym: Be-MaGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Praev. & Rehab. Sports medicine; Klinikum r. d. Isar; contact person: Mr. Johannes Scherr, MD
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2384/09
Record Dates: First submitted 2009-06-29; First posted 2009-07-07 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2009-07

CONDITIONS: Inflammation; Heart Failure; Sudden Cardiac Death
MeSH Terms: conditions — Inflammation; Heart Failure; Death, Sudden, Cardiac | interventions — Polyphenols; Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyphenols (non-alcoholic beer) (Active Comparator)
  Interventions: Dietary Supplement: polyphenols (non-alcoholic beer)
- beverage without polyphenols (Placebo Comparator)
  Interventions: Dietary Supplement: beverage without polyphenols

INTERVENTIONS:
Dietary Supplement: polyphenols (non-alcoholic beer) — 1.0 - 1.5 l non-alcoholic beer per day; 3 weeks before and during a marathon run
  Arms: polyphenols (non-alcoholic beer)
Dietary Supplement: beverage without polyphenols — 1.0 - 1.5 l of beverage without polyphenols (otherwise the same composition as non-alcoholic beer) per day; 3 weeks before and during a marathon run
  Arms: beverage without polyphenols

SUMMARY:
The purpose of the study is to determine the myocardial function and vascular adaptation after strenuous exercise in association with consumption of polyphenols. The investigators aim to investigate the effects of extreme endurance exercise on the inflammatory system. Furthermore, the role of the cardiovascular response and adaptive mechanisms of the vasculature are examined. Subclinical injuries to the myocardium and vascular wall are being investigated.

DETAILED DESCRIPTION:
Regular exercise leads to an improvement of cardiovascular risk factors in patients with coronary heart disease, atherosclerosis and metabolic disorders.

Aerobic exercise has anti-inflammatory effects. In contrast, the exertional exercise of marathon running causes an acute pro-inflammatory impulse. This may lead to myocardial injury and, in case of preexisting plaques, may result in plaque rupture and acute myocardial infarction.

We aim to define the critical role of inflammatory markers and cardiovascular risc factors as a predictor of an increased risk for myocardial and endothelial dysfunction in marathon runners.

Diagnostic tools include measurements of microvasculature, the large vessels and echocardiography. Inflammatory markers include high sensitive c-reactive protein (CRP) and interleukins.

All variations are analysed on the basis of consumption of polyphenols as they are found in in hops (Humulus lupus L.) and beer.

ELIGIBILITY:
Inclusion Criteria:

* men aged 20-60 years

Exclusion Criteria:

* manifested heart disease
* insulin dependent diabetes mellitus
* multi drug therapy
* GFR < 60 ml/min
* smokers
* neoplasia
* (former) alcoholism
* known malabsorption
* known chronic inflammatory disease

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker: Interleukin 6 and Interleukin 10 | pre-, post-, one & three day follow-up

SECONDARY OUTCOMES:
E/E' ratio | pre-, post-, one & three day follow-up
AV-ratio | pre-, post-, one & three day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prevention and Sports medicine, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Schoenfeld J, Schindler MJ, Haller B, Holdenrieder S, Nieman DC, Halle M, La Gerche A, Scherr J. Prospective long-term follow-up analysis of the cardiovascular system in marathon runners: study design of the Pro-MagIC study. BMJ Open Sport Exerc Med. 2020 Jul 19;6(1):e000786. doi: 10.1136/bmjsem-2020-000786. eCollection 2020. PMID 32704381
- [Derived] Roeh A, Schuster T, Jung P, Schneider J, Halle M, Scherr J. Two dimensional and real-time three dimensional ultrasound measurements of left ventricular diastolic function after marathon running: results from a substudy of the BeMaGIC trial. Int J Cardiovasc Imaging. 2019 Oct;35(10):1861-1869. doi: 10.1007/s10554-019-01634-5. Epub 2019 Jun 1. PMID 31154595
- [Derived] Scherr J, Halle M. Amendment on the findings of two previously published articles. Eur J Prev Cardiol. 2018 Mar;25(5):558. doi: 10.1177/2047487317754279. Epub 2018 Jan 26. No abstract available. PMID 29370708
- [Derived] Scherr J, Schuster T, Pressler A, Roeh A, Christle J, Wolfarth B, Halle M. Repolarization perturbation and hypomagnesemia after extreme exercise. Med Sci Sports Exerc. 2012 Sep;44(9):1637-43. doi: 10.1249/MSS.0b013e318258aaf4. PMID 22543737
- [Derived] Scherr J, Braun S, Schuster T, Hartmann C, Moehlenkamp S, Wolfarth B, Pressler A, Halle M. 72-h kinetics of high-sensitive troponin T and inflammatory markers after marathon. Med Sci Sports Exerc. 2011 Oct;43(10):1819-27. doi: 10.1249/MSS.0b013e31821b12eb. PMID 21448080